CLINICAL TRIAL: NCT01864863
Title: An Open-label, Randomized, Single-dose, 2-way Crossover Study to Compare the Pharmacokinetics of Traclear 62.5 mg 2 Tablets and HGP1206 125mg 1 Tablet in Healthy Male Volunteers
Brief Title: To Compare the Pharmacokinetics of Traclear 62.5 mg Tablets and HGP1206 125mg 1 Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-BOTAN-101
Record Dates: First submitted 2013-05-20; First posted 2013-05-30 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test→Reference (Experimental): HGP1206 125 mg 1 tablet → Traclear 62.5 mg 2 tablets
  Interventions: Drug: HGP1206; Drug: Traclear
- Reference→Test (Experimental): Traclear 62.5 mg 2 tablets → HGP1206 125 mg 1 tablet
  Interventions: Drug: HGP1206; Drug: Traclear

INTERVENTIONS:
Drug: HGP1206 — One Bosentan 125 mg tablet
  Other Names: Bosentan 125 mg
Drug: Traclear — Two Bosentan 62.5 mg tablets
  Other Names: Traclear 62.5 mg

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of two Traclear 62.5 mg tablets and one HGP1206 125 mg tablet in healthy male volunteers.

DETAILED DESCRIPTION:
An Open-label, Randomized, Single-dose, 2-way Crossover Study to Compare the Pharmacokinetics and safety of Traclear 62.5 mg Tablets and HGP1206 125mg Tablet in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age between 20 and 55
* Signed informed consent

Exclusion Criteria:

* Has a history of Primary pulmonary hypertension to investigational product ingredients
* Hypotension or hypertension

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
AUClast | 0-24h
Cmax | 0-24h

SECONDARY OUTCOMES:
Tmax | 0~24h
AUCinf | 0~24h
t1/2 | 0~24h

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No